CLINICAL TRIAL: NCT05265611
Title: Youth as Community Mental Health Workers in Humanitarian Settings: A Pilot Test of the Mechanisms of Effect on Their Own Well Being
Brief Title: Syrian Refugee Young Adults as Community Mental Health Workers-Lebanon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rema Afifi (Other)
Responsible Party: Sponsor-Investigator, Rema Afifi, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202107337
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Mental Health; Stress, Psychological
Keywords: Lebanon; Refugee; Problem Management Plus; RCT; Psychosocial intervention
MeSH Terms: conditions — Psychological Well-Being; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young Adult Community Mental Health Worker (Experimental): Syrian refugee young adults will be trained to implement Problem Management Plus (PM+): a WHO evidence-based low intensity mental health intervention to Syrian refugee adults in their community. They will complete 4 surveys to measure outcomes and mechanisms.
  Interventions: Behavioral: low intensity psychosocial intervention - Problem Management Plus (PM+)
- Young Adult Tutors (Active Comparator): Syrian refugee young adults will be trained to tutor elementary school students in their community.They will complete 4 surveys to measure outcomes and mechanisms.
  Interventions: Behavioral: Tutoring
- Young Adut Control Group (No Intervention): Syrian refugee young adults in the control group will only complete the surveys. They will complete 4 surveys to measure outcomes and mechanisms.

INTERVENTIONS:
Behavioral: low intensity psychosocial intervention - Problem Management Plus (PM+) — Syrian refugee young adults will be trained to implement Problem Management Plus (PM+). PM+ is a low-intensity mental health intervention, developed by WHO, and delivered by non-specialized CMHW. It is a transdiagnostic treatment approach that includes four evidence-based problem solving and behavioral treatment techniques: managing stress, managing problems, get going/get doing, and social support. These strategies are implemented over five weekly sessions, of 90 minutes each.
  Arms: Young Adult Community Mental Health Worker
Behavioral: Tutoring — Young adults will be trained to tutor students in elementary school.
  Arms: Young Adult Tutors

SUMMARY:
In this pilot study, we aim to evaluate the feasibility, acceptability and fidelity of Syrian refugee young adults as community mental health workers (Y-CMHW), and the impact of this work on outcomes of wellbeing, coping and stress. In addition, we aim to assess the mechanisms leading to any changes in these outcomes.

DETAILED DESCRIPTION:
Involving youth and young adults (YYA) in work that impacts their communities has positive outcomes for youth wellbeing; and for their communities. But, YYA are often marginalized, particularly in humanitarian settings. YYA wellbeing is linked to seven key protective factors: positive emotions, hope, relationships, meaning, accomplishments, autonomy, and engagement. Understanding protective factors as potential mechanisms for intervention-related change in wellbeing is a priority for research in humanitarian settings.

Humanitarian crises increase mental health disorders; and 'normal' distress and psychological reactions affect a large percentage of the population. Yet, human resources for health are often insufficient to meet needs. Understanding the capacities of YYA to support communities in the context of disasters has been noted as a research imperative. Globally, task-sharing interventions train non-professional lay community members to provide mental health care. As one example, Problem Management Plus (PM+) trains community mental health workers (CMHW) and is effective in humanitarian settings for common mental disorders and other problems that emerge in response to crises.

The investigators propose to engage Syrian refugee young adults (YA) - aged 18-24 years, as YA CMHW, to implement PM+ with at-risk adults (18+ years) in their communities. The Syrian refugee crises, one of the worst humanitarian crises in recent history, provides a relevant setting to implement this project. Lebanon hosts ~1.5 million Syrian refugees, and about 60% of Syrian refugees aged 15-24 years are not employed, and not in school. The Specific Aims are:

Aim 1: Assess the effectiveness of being a YA-CMHW on their wellbeing, coping, and stress levels; as compared to (i) an active comparator group of Syrian refugee peers providing tutoring services; and (ii) a group of Syrian refugee peers that receives no intervention.

Aim 2: Identify the mechanisms associated with changes in wellbeing, coping, and stress. The conceptual model describes links between the intervention, the mechanisms, and outcomes.

Aim 3: Evaluate the feasibility, acceptability and fidelity of Syrian refugee YA as CMHW implementing PM+ with clients.

Results will (a) elucidate critical mechanisms through which engagement of YYA to support their community enhances their own wellbeing; (b) inform research around humanitarian/refugee settings, mental health, and Y-CMHW interventions; and (c) provide a robust basis for a follow-up study via a larger RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Syrian refugee
2. 18-24 years
3. have completed high school
4. at the time of screening, live in one of the 3 catchment areas of the field-based NGO partner (MAPs) in the Bekaa region of Lebanon
5. have been involved in NGOs or service to their community'
6. motivation to be a Community Mental Health Worker

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Wellbeing | Year 2 month 8- Year 4 month 8
  Self report through survey
Stress | Year 2 month 8 - Year 4 month 8
  Self report through survey and Hair Cortisol
Coping/Resilience | Year 2 month 8 - Year 4 month 8
  Self report through survey

SECONDARY OUTCOMES:
Mechanism-Positive emotions | Year 2 month 8 - Year 4 month 8
  Self report through survey
Mechanism-Supportive relationships | Year 2 month 8 - Year 4 month 8
  Self report through survey
Mechanism-Engagement | Year 2 month 8 - Year 4 month 8
  Self report through survey
Mechanism-Accomplishments | Year 2 month 8 - Year 4 month 8
  Self report through survey
Mechanism-Optimism/Hope | Year 2 month 8 - Year 4 month 8
  Self report through survey
Mechanism-Meaning/Purpose in life | Year 2 month 8 - Year 4 month 8
  Self report through survey
Mechanism-Control/Autonomy | Year 2 month 8 - Year 4 month 8
  Self report through survey

CONTACTS AND LOCATIONS:
Overall Officials: Rima A Afifi, PhD, Principal Investigator — University of Iowa College of Public Health
Locations (1):
- American University of Beirut, Faculty of Health Sciences, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlie results reported in publications will be shared with researchers.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months after article publication.
Access Criteria: "Access to trial IPD can be requested by researchers conducting independent scientific research, and will be provided following review and approval of a research proposal and analysis plan and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the Principal Investigator."

REFERENCES:
- [Result] Nakkash R, Ghandour L, Brown G, Panter-Brick C, Bomar H, Tleis M, Al Masri H, Fares M, Al Halabi F, Najjar Y, Louis B, Hodroj M, Chamoun Y, Zarzour M, Afifi RA. Syrian refugee young adults as community mental health workers implementing problem management plus: Protocol for a pilot randomized controlled trial to measure the mechanisms of effect on their own wellbeing, stress and coping. Contemp Clin Trials Commun. 2024 Jun 28;40:101325. doi: 10.1016/j.conctc.2024.101325. eCollection 2024 Aug. PMID 39045391
- [Result] Ghandour L, Brown G, Tleis M, Al Masri H, Fares M, Al Halabi F, Najjar Y, Louis B, Afifi RA, Nakkash R. Structural and political determinants of health among Syrian refugee young adults in the Bekaa, Lebanon: a prospective cohort study of the impact of security raids on perceived discrimination and well-being. BMJ Open. 2024 Dec 5;14(12):e087777. doi: 10.1136/bmjopen-2024-087777. PMID 39638591
- [Result] Nakkash R, Fares M, Tleis M, Mugharbil A, Antaby M, Al Masri H, Ghandour L, Al Halabi F, Najjar Y, Louis B, Afifi RA. (2024). Power Sharing in Community-Engaged Research with Syrian Refugees in Lebanon: Using community engagement to shape Intervention Fit to Context. Social Science and Medicine, Mental Health; 6(4): 100358, https://doi.org/10.1016/j.ssmmh.2024.100358.